CLINICAL TRIAL: NCT02318433
Title: Intra-Articular Dexamethasone to Prevent Post-Traumatic Osteoarthritis: A Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sanjeev (Sanj) Kakar, M.D., M.B.A., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 14-004033
Record Dates: First submitted 2014-12-08; First posted 2014-12-17 (Estimated); Last update posted 2020-04-13 (Actual); Status verified 2020-03

CONDITIONS: Distal Radius Fracture; Osteoarthritis
Keywords: DRF; PTOA; dexamethasone
MeSH Terms: conditions — Wrist Fractures; Osteoarthritis | interventions — Dexamethasone; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Experimental): Subjects receive dexamethasone (4 mg) injection within the radiocarpal joint either in clinic or in the OR.
  Interventions: Drug: Dexamethasone
- Saline (Placebo Comparator): Subjects receive sterile saline (4 mg) injection within the radiocarpal joint either in clinic or in the OR.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexamethasone — Data demonstrates that low doses of dexamethasone preserves chondrocyte viability, protects collagen, and maintains proteoglycan synthesis in cartilage subjected to injurious compression.
  Arms: Dexamethasone
Drug: Saline
  Arms: Saline

SUMMARY:
The primary aim of the study is to see if a single wrist injection (intra-articular) of dexamethasone at the time of treatment will reduce the incidence of early-onset of post traumatic osteoarthritis.

DETAILED DESCRIPTION:
Our hypothesis is that the intra-articular administration of dexamethasone soon after joint injury will prevent the subsequent development of PTOA, and restore normal joint homeostasis. We plan to generate the data needed to test this hypothesis in a Phase 0 (pilot) clinical trial using patients who have suffered distal radius fractures.

ELIGIBILITY:
Inclusion Criteria:

1. Unstable distal radius fracture
2. Fracture type AO B1, B2, B3, C1, C2 or C3.
3. 18-65 years old
4. Understand and read English
5. Community dwelling (not in assisted living or NH)

Exclusion criteria:

1. Open or bilateral DRF
2. Associated upper extremity carpal fracture or carpal ligament injuries requiring casting or surgical repair at the time of DRF fixation.
3. Greater than 2 weeks post injury
4. Neurologic disorders affecting the hand, wrist or arm.
5. History of permanent dementia, Alzheimer's or other neurologic dx
6. Substance abuse
7. Pathologic fractures
8. Known pregnancy
9. Radiocarpal joint arthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-12; Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

PRIMARY OUTCOMES:
PTOA incidence | 3 years
  Primary outcome measure will incidence of post-traumatic osteoarthritis, determined by joint space narrowing, as measured radiologically.

SECONDARY OUTCOMES:
Functional assessment | 3 years
  A composite of clinical measurements of grip strength and pinch strength.
Patient-rated evaluations | 3 years
  Composite scores from patient-rated evaluations including the Disabilities of the Arm Shoulder and Hand (DASH), the Michigan Hand Questionnaire (MHQ), and the Patient-Rated Wrist Evaluation (PRWE).

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Kakar, M.D., M.B.A, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials